CLINICAL TRIAL: NCT05950126
Title: Is Pain Perception Communicated Through Mothers? Maternal Pain Catastrophizing Score is Related With Children's Postoperative Circumcision Pain
Brief Title: Maternal Pain Catastrophizing Score is Related With Children's Postoperative Circumcision Pain
Status: Completed | Type: Observational
Sponsor: Sevda Akdeniz,MD (Other)
Responsible Party: Sponsor-Investigator, Sevda Akdeniz,MD, Samsun University, Samsun University
Organization: Samsun University (Other)
Other Study IDs: B.30.2.ODM.0.20.08/80-165
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Pain Catastrophizing
Keywords: postoperative pain; circumcision; pain catastrophizing; mother; children; VAS
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: low pain catastrophizing score in mother
  Interventions: Other: pain catastrophizing scala
- Group 2: high pain catastrophizing score in mother
  Interventions: Other: pain catastrophizing scala

INTERVENTIONS:
Other: pain catastrophizing scala — The PCS, a 13-item self-report inventory used to determine the extent to which individuals catastrophize in response to pain, was developed. Total possible scores range from 0 to 52, with higher scores indicating negative results.
  The Turkish version was tested for reliability and validity and the Cronbach alpha coefficient was measured at 0.90. PCS scores of 16 or lower are regarded as normal, and scores of 17 or above as high.

SUMMARY:
The aim of this study was to evaluate the relation of maternal pain catastrophizing score with child's who underwent circumcision postoperative pain. A cross-sectional study and this study was performed at the Samsun University, Samsun Training and Research Hospital, Samsun, Türkiye. The mothers were divided into low pain catastrophizing (Group 1) and high pain catastrophizing (Group 2) group. Children's postoperative pain intensity was measured using the visual analog scale (VAS) and a faces pain scale (FPS).

DETAILED DESCRIPTION:
Now, the study is continuing.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-12 years,
* Being operated under general anesthesia.

Exclusion Criteria:

* Children without biological mothers, or with a parent other than the mother,
* Children aged under five or over 12,
* History of previous surgery,
* Being operated under regional anesthesia,
* Use of analgesic, antiepileptic, or sedative medications, and
* Other procedures being performed in addition to circumcision (such as herniorrhaphy, tonsillectomy, orchiopexy, and appendectomy).

Ages: 5 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Among the children who come to the preoperative anesthesia outpatient clinic with their mothers to undergo elective circumcision will be accepted if their mothers will be agreed to participate in the study. Volunteer mothers at the anesthesia outpatient clinic will be given a questionnaire to fill out and provided informed consent.
Study Population: Among the children who come to the preoperative anesthesia outpatient clinic with their mothers to undergo elective circumcision will be accepted if their mothers agreed to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
PCS, mother, and child | 18 month
  Authors will be investigated the relationship between maternal pain catastrophizing score levels and the postoperative pain experienced by the child. Empathy towards pain is necessary to notice, understand, and respond to another person's pain. Children develop empathy towards pain over time, which may be related to social learning.
  Pain Catastrophizing scale (PCS): The PCS is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale, from 0 (not at all) to 4 (always), people are asked to rate how often they experience the mentioned thoughts and feelings when they are in pain. The overall score has a range of 0-52.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Suren M, Okan I, Gokbakan AM, Kaya Z, Erkorkmaz U, Arici S, Karaman S, Kahveci M. Factors associated with the pain catastrophizing scale and validation in a sample of the Turkish population. Turk J Med Sci. 2014;44(1):104-8. doi: 10.3906/sag-1206-67. PMID 25558568
- See also: Reference article — http://pubmed.ncbi.nlm.nih.gov/25558568/